CLINICAL TRIAL: NCT04867148
Title: The Prediction and Prevention of Disease by Using Big Data in Motion Analysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Lee Jung Sub, Professor, Pusan National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PNUH orthopaedics
Record Dates: First submitted 2021-04-27; First posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Ankylosing Spondylitis; Adolescent Idiopathic Scoliosis; Gait Analysis
Keywords: Gait analysis; Spine
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gait analysis (Experimental): Gait analysis of patients with ankylosing spondylitis, patients with adoldescent idiopathic scoliosis and control group.
  Interventions: Device: Inertial measurement unit sensor-based gait analysis system

INTERVENTIONS:
Device: Inertial measurement unit sensor-based gait analysis system — Gait analysis was performed on 20-m long corridor to collect gait data on more than 23 strides. The gait protocol was performed with an IMU sensor-based gait analysis system (DynaStab™, JEIOS, South Korea) consisting of a shoe-type data logger (Smart Balance1 SB-1, JEIOS, South Korea) and a data acquisition system (DynaStab-Spotfire1, Tibco Spotfire 7.10). The shoe-type data logger included an IMU sensor (IMU-3000™, InvenSense, USA) that measured tri-axial acceleration (up to ± 6 g) and tri-axial angular 136 velocity (up to ± 500˚ s-1) along three orthogonal axes.12,16 The IMU sensors were installed in both shoe outsoles, and the data were transmitted wirelessly to a data acquisition system via Bluetooth®. Shoe sizes were adapted to each participant, with available sizes ranging from 225 mm to 280 mm. The local coordinate system for the IMU sensors included the 140 anteroposterior, mediolateral, and vertical directions.

SUMMARY:
Variable patterns of gait disturbance can be found in patients with spine disease including the problems of gait initiation, freezing of gait, reduced balance and postural control, reduced step lengths, increased step times, and slow walking speed.

ELIGIBILITY:
Inclusion Criteria:

* Pusan National University Hospital orthopedics, otorhinolaryngology, neurology outpatient or inpatient who agreed to the study.
* For adult men and women 18 years of age or older.

Exclusion Criteria:

* Patients unable to walk independently.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
gait asymmetry | for 1minute walking
  comparing the swing times performed by one leg with respect to the swing times performed by the other, according to the following formula: GA = 100 x ln(SSWT/LSWT)

CONTACTS AND LOCATIONS:
Overall Officials: jungsub Lee, M.D., Ph.D., Study Chair — Pusan National University Hospital
Locations (1):
- Pusan National University Hospital, Busan, Seo-gu, South Korea